CLINICAL TRIAL: NCT04485611
Title: Prehabilitation of Veterans With Exercise and Nutrition (PREVENT)
Brief Title: Prehabilitation of Veterans With Exercise and Nutrition
Acronym: PREVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F3468-P; 728745 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2020-07-02; First posted 2020-07-24 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Frailty
Keywords: frailty; exercise training; telemedicine; nutritional support
MeSH Terms: conditions — Frailty | interventions — Resistance Training; Nutritional Support

STUDY DESIGN:
Intervention Model Description: The intervention will consist of a period of supervised multimodal prehabilitation prior to high-risk surgery (aerobic and resistance training sessions 3 times/week plus nutritional support) delivered using telehealth technology, and similar sessions resuming after surgery and for up to 6 weeks (rehabilitation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prehabilitation (Experimental): This pilot cohort will undergo an intervention and will be followed for up to 6 months. The study does not include a comparator group.
  Interventions: Behavioral: Supervised aerobic + resistance training and nutritional support

INTERVENTIONS:
Behavioral: Supervised aerobic + resistance training and nutritional support — The intervention will consist of individualized exercise training delivered remotely using VA telehealth technology, combined with nutritional support consisting of tailored nutritional advice, protein supplementation, multivitamin and vitamin D supplements]]. Adherence to the intervention will be enhanced by use of automated text messages and monitored using activity trackers.
  Other Names: Multimodal prehabilitation

SUMMARY:
The goal of VA's RR&D office is to maximize functional recovery. This proposal will allow the investigators to test an intervention that combines the fundamentals of Physical Medicine and Rehabilitation with state-of-the-art nutritional support and innovations in care such as telehealth and the use of activity trackers to optimize patients before high-risk surgery. This intervention has the potential to not only reduce complications and hospital readmissions, but also to maximize functional recovery and quality of life for thousands of Veterans undergoing high-risk surgery every year. Furthermore, the proposal is the first step in the design and implementation of prehabilitative services for Veterans living in rural areas and those with inadequate support or transportation.

DETAILED DESCRIPTION:
Approximately half a million operations are performed each year in VA hospitals across the country. Veterans undergoing high-risk surgery have a 1 in 5 chance of suffering complications, a 1 in 10 chance of being readmitted to the hospital within 30 days, and a 1 in 50 chance of dying within 30 days. Long-term survival is significantly reduced for those patients who have perioperative complications, even if they survive to leave the hospital.

Low fitness and poor functional status are among the strongest predictors of postsurgical complications. Prehabilitation takes advantage of the weeks leading up to surgery in order to improve fitness, mobility and nutrition in preparation for the upcoming surgical stress. Indeed, prehabilitation has been shown to improve fitness and reduce complications and quality of life in high-risk surgical patients. The most effective prehabilitation programs combine exercise plus nutritional support (are multimodal), and provide exercise that is supervised and individualized, ensuring the appropriate exercise intensity and increasing it gradually according to improvements in fitness and strength. Most supervised prehabilitation programs are facility-based, but travel time, distance, and transportation limit participation. Unfortunately, home-based prehabilitation programs have shown small effect sizes and low compliance rates, likely because adequate training intensity is required in programs of such short duration, which is often not achieved with unsupervised home-based programs. A prehabilitation program that is delivered using telehealth would be ideal, because it combines accessibility with supervision, encouraging compliance and ensuring adequate training intensity, but such programs do not currently exit within the VA.

The investigators aim to determine the feasibility, acceptability, safety, and effect size estimates for outcomes of interest of a short-term (3-4 week) multimodal prehabilitation intervention that is supervised and individualized, yet is delivered at home using telehealth technology. The exercise program will consist of 3 days of supervised telehealth exercise sessions per week consisting of moderate intensity aerobic training and resistive and functional training. Nutritional support will consist of tailored nutritional advice, whey protein supplementation and multivitamin and vitamin D supplementation during prehabilitation and following hospital discharge for 6 weeks. Compliance with the interventions will be enhanced by daily automated text messages using the VA Annie App. In addition, participants will be contacted weekly in order to identify problems with compliance and to provide counseling. Post-operative exercise sessions will resume as early as 1 week postoperatively and progressed as allowed according to the type of surgery. Text messages and weekly calls will also resume postoperatively until the 6-week follow-up visit to encourage progressive increases in unsupervised physical activity and nutritional support. Objective physical activity data will be collected using physical activity trackers, which patients will wear from the time of enrollment until the 6-week postoperative follow-up visit. Follow-up will continue for a total of 6 months postoperatively.

The main outcomes of interest include feasibility (acceptance rates), acceptability (compliance rates), and safety (number of adverse events). The investigators will also measure changes in fitness, nutritional state, anxiety and depression, and health-related quality of life throughout the study period in order to estimate effect sizes, which will inform a future randomized trial. The proposed work combines several innovations in the delivery of exercise and nutrition and applies them to the perioperative high-risk population for the first time. It constitutes the first step toward the study of a multimodal "tele-prehabilitation" program on postoperative and long-term outcomes following high-risk surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for high-risk surgery
* Time from assessment to surgery 21 days
* Age 50 years
* English speaking
* 5RSTS time >11 sec and/or TMST score 25% percentile for gender/age

Exclusion Criteria:

* A score of <21 (high school) or <20 (less than high school) on the Montreal Cognitive Assessment (MoCA)
* Dementia diagnosis
* Inability to complete physical function assessment
* ASA categories 4 and 5
* Living in skilled nursing facility
* No access to a telephone
* Advanced chronic kidney disease (KDIGO stage 4 and 5)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atilio Barbeito, MD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 05/27/2021 Recruitment ended 10/18/2023
Pre-assignment Details: 20 patients were enrolled in the study. One patient underwent the baseline evaluation but withdrew before starting the intervention.
  One patient enrolled but his clinical condition changed and was therefore withdrawn from the study before the initial baseline evaluation was completed.
  A total of 18 participants started the prehabilitation intervention.
Groups:
- Overall Study: This pilot cohort will undergo an intervention and will be followed for up to 6 months. The study does not include a comparator group.
  Supervised aerobic + resistance training and nutritional support: The intervention will consist of individualized exercise training delivered remotely using VA telehealth technology, combined with nutritional support consisting of tailored nutritional advice, protein supplementation, multivitamin and vitamin D supplements]]. Adherence to the intervention will be enhanced by use of automated text messages and monitored using activity trackers.
Period: Prehabilitation
Arm/Group | Overall Study
Started | 18
Completed | 17 (One patient enrolled and began the prehabilitation intervention but his clinical condition changed and was deemed ineligible fo surgery, and was therefore withdrawn from the study.)
Not Completed | 1
Not completed — Physician Decision | 1
Period: Rehabilitation
Arm/Group | Overall Study
Started | 14 (17 patients completed the prehabilitation intervention. Three patients withdrew from the study after surgery and before starting the rehabilitation phase.)
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 63 patients were screened and offered to participate, and 29 agreed to enroll and undergo a physical function evaluation. Of these, 20 patients (69%) were frail or pre-frail and qualified for the intervention. One patient withdrew before the initial evaluation was completed. One patient completed the baseline evaluation but was later withdrawn from the study due to a change in his medical condition.
Groups:
- Prehabilitation: This pilot cohort will undergo an intervention and will be followed for up to 6 months. The study does not include a comparator group.
  Supervised aerobic + resistance training and nutritional support: The intervention will consist of individualized exercise training delivered remotely using VA telehealth technology, combined with nutritional support consisting of tailored nutritional advice, protein supplementation, multivitamin and vitamin D supplements. Adherence to the intervention will be enhanced by use of automated text messages and monitored using activity trackers.
Arm/Group | Prehabilitation
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 63.95 [50 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 30.29 [19.8 to 37.3]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility, Measured as Acceptance Rate
Description: Acceptance rate will be calculated as the number of enrolled divided by the number of eligible patients.
Time Frame: From initial screening to enrollment (~7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Prehabilitation
Number analyzed (Participants) | 29
Participants | 20

2. Primary Outcome: Acceptability, Measured as Compliance Rate
Description: For the exercise intervention, the investigators will measure the percentage of patients completing 75% of sessions divided by the number of enrolled patients. For the nutritional intervention, compliance will be measured by the percentage of patients with 75% adherence to protein intake goal, as assessed using the text message-based nutrition diary and 24-hour recall administered during the weekly telephone call.
Time Frame: End of prehabilitation (week 3) and end of rehabilitation (week 14)
Population: 20 patients were enrolled in the study. Two patients withdrew before starting the intervention and one patient began the prehabilitation phase but had to be withdrawn due to progression of disease. Two patients withdrew after recovering from surgery and before starting the rehabilitation phase. The last patient in the cohort was not offered rehabilitation (funding ended). A total of 14 patients began the rehabilitation phase of the intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Study: This cohort underwent supervised aerobic + resistance training and nutritional support. The intervention consisted of individualized exercise training delivered remotely using VA telehealth technology 3 times per week during the 3 weeks leading up to surgery, combined with nutritional support consisting of tailored nutritional advice, protein supplementation, multivitamin and vitamin D supplements. Adherence to the intervention was enhanced by use of automated text messages.
  The study did not include a comparator group.
Arm/Group | Study
Number analyzed (Participants) | 20
Participants
  Prehabilitation -Exercise | 16
  Rehabilitation - Exercise: number analyzed (Participants) | 14
  Rehabilitation - Exercise | 11
  Prehabilitation - Nutrition | 12
  Rehabilitation - Nutrition: number analyzed (Participants) | 14
  Rehabilitation - Nutrition | 6

3. Primary Outcome: Safety, Measured as the Number of Adverse Events During Exercise.
Description: A significant injury or medical event is defined as an event that causes the participant to seek attention from a health professional or limits their activities of daily living for at least two days.
Time Frame: Throughout the study period, and summarized at the end of prehabilitation (week 3) and end of rehabilitation (week 14)
Measure: Number; unit: participants
Arm/Group | Prehabilitation
Number analyzed (Participants) | 18
participants | 0

4. Secondary Outcome: Physical Function - Aerobic Endurance
Description: Aerobic endurance will be assessed using the 2-minute step test (2MST). The 2MST requires that tested individuals march in place as fast as possible for 2 minutes while lifting the knees to a height midway between their patella and iliac crest when standing (typically marked on the wall using tape). Scoring involves counting the number of times the right knee reaches the tape level in two minutes and comparing against normative values for age. A higher number denotes better aerobic endurance.
Time Frame: Baseline, end of prehabilitation (week 3), post-surgery (variable but ~week 8), and post-rehabilitation (week 14)
Measure: Mean (Standard Deviation); unit: Step Count
Groups:
- Baseline; Post-prehabilitation: This cohort underwent supervised aerobic + resistance training and nutritional support. The intervention consisted of individualized exercise training delivered remotely using VA telehealth technology 3 times per week during the 3 weeks leading up to surgery, combined with nutritional support consisting of tailored nutritional advice, protein supplementation, multivitamin and vitamin D supplements. Adherence to the intervention was enhanced by use of automated text messages.
  The study did not include a comparator group.
- Post-surgery; Post-rehabilitation: This cohort underwent supervised aerobic + resistance training and nutritional support. The intervention consisted of individualized exercise training delivered remotely using VA telehealth technology 3 times per week during the 6 weeks following recovery from surgery, combined with nutritional support consisting of tailored nutritional advice, protein supplementation, multivitamin and vitamin D supplements. Adherence to the intervention was enhanced by use of automated text messages.
  The study did not include a comparator group.
Arm/Group | Baseline | Post-prehabilitation | Post-surgery | Post-rehabilitation
Number analyzed (Participants) | 18 | 18 | 14 | 14
Step Count | 79.11 (19.73) | 105.41 (25.15) | 86.73 (16.21) | 115.38 (21.85)

5. Secondary Outcome: Physical Function - Lower Extremity Strength and Balance
Description: Lower extremity strength and balance will be assessed using the 5-repetition sit-to-stand test (5XSST). The 5XSST assesses functional lower extremity strength, transitional movements, balance, and fall risk in older adults. The 5XSST scoring is based on the amount of time (to the nearest decimal in seconds) a patient is able to transfer from a seated to a standing position and back to sitting five times. The lower the time to complete the test the better the outcome of the test. The age matched norms score are 11.4 seconds for 60-69 years age groups and 12.6 seconds and 14.8 seconds for 70-79 and 80-89 years of age group ,respectively.
Time Frame: Baseline, end of prehabilitation (week 3), post-surgery (variable but typically ~week 8), and post-rehabilitation (week 14)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Baseline | Post-prehabilitation | Post-surgery | Post-rehabilitation
Number analyzed (Participants) | 18 | 18 | 14 | 14
seconds | 14.47 (4.61) | 9.93 (2.14) | 11.37 (2.62) | 8.85 (1.49)

6. Secondary Outcome: Hospital Anxiety & Depression Scale (HADS): Anxiety (HADS-A)
Description: Pre to post intervention changes in anxiety and depression as measured by the Hospital Anxiety & Depression Scale (HADS) questionnaire. Lower scores are better.
  0-7: Indicates no or minimal anxiety. 8-10: Suggests mild anxiety. 11-15: Indicates moderate anxiety. 16-21: Suggests severe anxiety.
Time Frame: Baseline, end of prehabilitation (week 3), post-surgery (variable but ~week 8), post-rehabilitation (week 14), and 4-month post-rehabilitation follow-up (week 32)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 32-week Follow-up: This is a follow-up assessment 18 weeks following the end of the rehabilitation intervention
Arm/Group | Baseline | Post-prehabilitation | Post-surgery | Post-rehabilitation | 32-week Follow-up
Number analyzed (Participants) | 19 | 17 | 14 | 14 | 14
units on a scale | 5.21 (3.71) | 4.23 (2.97) | 4.21 (2.61) | 2.92 (2.87) | 4.21 (4.17)

7. Secondary Outcome: Hospital Anxiety & Depression Scale (HADS): Depression (HADS-D)
Description: Pre to post intervention changes in anxiety and depression as measured by the Hospital Anxiety & Depression Scale (HADS) questionnaire. Lower scores are better.
  0-7: Indicates no or minimal depression. 8-10: Suggests mild depression. 11-15: Indicates moderate depression. 16-21: Suggests severe depression.
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | Post-prehabilitation | Post-surgery | Post-rehabilitation | 32-week Follow-up
Number analyzed (Participants) | 19 | 17 | 14 | 14 | 14
units on a scale | 3.16 (2.83) | 2.71 (1.93) | 3.57 (2.85) | 1.77 (1.92) | 3.57 (4.41)

8. Secondary Outcome: Short Form 36 (SF-36)
Description: Pre to post intervention changes in quality of life as measured by the Short Form 36 (SF-36) questionnaire.
  The SF-36 is a 36-item patient-reported questionnaire designed to assess health-related quality of life. Scores range from 0 to 100, with higher scores indicating better health.
Time Frame: Baseline, post-rehabilitation (~week 14), and 4-month post-rehabilitation follow-up (week 32)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Post-rehabilitation | 32-week Follow-up
Number analyzed (Participants) | 19 | 14 | 14
score on a scale | 69.04 (17.48) | 74.60 (16.41) | 68.21 (15.74)

ADVERSE EVENTS:
Time Frame: Adverse events were captured throughout the study period and summarized at the end of prehabilitation (week 3) and end of rehabilitation (week 14)
Arm/Group | Baseline | Post-prehabilitation | Post-surgery | Post-rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
The data used to calculate the effect of the interventions was derived from in-person assessments when available. Due to the nature of the study, some assessments could not be completed in person and were completed using telehealth technology.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT04485611/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT04485611/ICF_000.pdf